CLINICAL TRIAL: NCT05725967
Title: Endoscopic Metabolic and Bariatric Therapies
Acronym: EMBTs
Status: Enrolling by invitation | Type: Observational
Sponsor: Christopher C. Thompson, MD, MSc (Other)
Responsible Party: Sponsor-Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Other Study IDs: 2022P001757
Record Dates: First submitted 2022-12-29; First posted 2023-02-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Obesity, Morbid; Obesity Associated Disorder; Bariatric Surgery Candidate; Fistula, Gastric; Roux-en-y Anastomosis Site; Ulcer, Gastric; Abdominal Pain; Abdominal Obesity; Complication of Surgical Procedure; Complication of Treatment; Complication,Postoperative; Weight Gain; Weight Loss; Leak, Anastomotic; Delayed Gastric Emptying Following Procedure
Keywords: Roux-en-Y Gastric Bypass; Sleeve Gastrectomy; laparoscopic adjustable gastric banding; gastroplasty with endoscopic myotomy (GEM); endoscopic sleeve gastroplasty (ESG); transoral outlet reduction (TORe); primary obesity surgery endoluminal (POSE); restorative obesity surgery endoluminal (ROSE); intragastric balloons (IGB); aspiration therapy; pylorus sparing antral myotomy (PSAM); gastric emptying breath test (GEBT)
MeSH Terms: conditions — Obesity; Obesity, Morbid; Gastric Fistula; Stomach Ulcer; Abdominal Pain; Obesity, Abdominal; Postoperative Complications; Weight Gain; Weight Loss; Anastomotic Leak | interventions — immunoglobulin B; Bariatric Surgery; Argon Plasma Coagulation; Gastroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Obesity Endoscopic Procedures: Primary endoscopic procedures for treatment of obesity.
  Interventions: Procedure: Primary Obesity Endoscopic Procedures; Device: Endoscopic Sleeve Gastroplasty, Trans-oral Outlet Reduction; Device: Intragastric Balloon; Device: Primary obesity surgery endoluminal, Restorative obesity surgery endoluminal; Device: Argon Plasma Coagulation, Gastroplasty with Endoscopic Myotomy, Bariatric Endoscopic Antral Myotomy, Pylorus Sparing Antral Myotomy; Device: Aspiration Therapy
- Endoscopic Revision of Bariatric Surgical Procedures: Endoscopic revision of post-bariatric surgical complications.
  Interventions: Procedure: Endoscopic Revision of Bariatric Surgical Procedures; Device: Endoscopic Sleeve Gastroplasty, Trans-oral Outlet Reduction; Device: Primary obesity surgery endoluminal, Restorative obesity surgery endoluminal; Device: Argon Plasma Coagulation, Gastroplasty with Endoscopic Myotomy, Bariatric Endoscopic Antral Myotomy, Pylorus Sparing Antral Myotomy
- Bariatric Surgery Procedures: Bariatric surgical procedures.
  Interventions: Procedure: Bariatric Surgery Procedures

INTERVENTIONS:
Procedure: Primary Obesity Endoscopic Procedures — Any primary endoscopic procedure for treatment of obesity including endoscopic sleeve gastroplasty (ESG), intragastric balloons (IGB), Aspiration therapy, pylorus sparing antral myotomy (PSAM), primary obesity surgery endoluminal (POSE), gastroplasty with endoscopic myotomy (GEM).
  Other Names: ESG, Aspiration Therapy, IGB, POSE, GEM, PSAM, BEAM, EMBTs
  Groups: Primary Obesity Endoscopic Procedures
Procedure: Endoscopic Revision of Bariatric Surgical Procedures — Any endoscopic revision procedure in a post-bariatric surgical patient, including transoral outlet reduction (TORe), restorative obesity surgery endoluminal (ROSE), argon plasma coagulation of the outlet (APC), endoscopic suturing.
  Other Names: TORe, ROSE, APC
  Groups: Endoscopic Revision of Bariatric Surgical Procedures
Procedure: Bariatric Surgery Procedures — Any bariatric surgical procedure including Roux-en-Y gastric bypass (RYGB), laparoscopic sleeve gastroplasty (LSG), laparoscopic adjustable gastric banding (LAGB)
  Other Names: RYGB, LSG, LAGB
  Groups: Bariatric Surgery Procedures
Device: Endoscopic Sleeve Gastroplasty, Trans-oral Outlet Reduction — Any endoscopic procedure using an endoscopic suturing device for primary obesity treatment or revision of post bariatric complications.
  Other Names: ESG, TORe
  Groups: Endoscopic Revision of Bariatric Surgical Procedures; Primary Obesity Endoscopic Procedures
Device: Intragastric Balloon — An endoscopic bariatric procedure involving the placement of an intragastric balloon.
  Other Names: IGB
  Groups: Primary Obesity Endoscopic Procedures
Device: Primary obesity surgery endoluminal, Restorative obesity surgery endoluminal — Any endoscopic procedure using an endoscopic plicating device for primary obesity treatment or revision of post bariatric complications.
  Other Names: POSE, ROSE
  Groups: Endoscopic Revision of Bariatric Surgical Procedures; Primary Obesity Endoscopic Procedures
Device: Argon Plasma Coagulation, Gastroplasty with Endoscopic Myotomy, Bariatric Endoscopic Antral Myotomy, Pylorus Sparing Antral Myotomy — Electrosurgical interventions for obesity. Use of electrosurgical devices, such as electrocautery for the primary treatment of obesity or obesity related complications.
  Other Names: APC, GEM, BEAM, PSAM
  Groups: Endoscopic Revision of Bariatric Surgical Procedures; Primary Obesity Endoscopic Procedures
Device: Aspiration Therapy — Placement of an aspiration therapy device for the treatment of obesity.
  Other Names: Aspire
  Groups: Primary Obesity Endoscopic Procedures

SUMMARY:
This is a prospective collection of data from adult patients who have had an endoscopic metabolic and bariatric endoscopy procedure (EMBT) for primary or revision surgical procedures for obesity.

DETAILED DESCRIPTION:
The Investigators will be collecting data on bariatric patients post-bariatric surgery, post-endoscopic revision of bariatric surgical complications and post-endoscopic metabolic and bariatric therapies (including but not limited to roux-en-y gastric bypass, sleeve gastrectomy, laparoscopic adjustable gastric banding, gastroplasty with endoscopic myotomy (GEM), endoscopic sleeve gastroplasty (ESG), transoral outlet reduction (TORe), primary obesity surgery endoluminal (POSE), restorative obesity surgery endoluminal (ROSE), intragastric balloons (IGB), aspiration therapy and pylorus sparing antral myotomy) to review demographics, adverse events, medications, radiology, procedure time, cost, comorbidity resolution and resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* patients from Mass General Brigham
* any patient having an endoscopic primary obesity procedure
* any patient having an endoscopic post-bariatric surgical revision procedure
* any patient having a bariatric surgical procedure

Exclusion Criteria:

* patients without past surgical and medical history medical records in the Mass General Brigham system
* patients unwilling to allow for medical record review at Mass General Brigham

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients registered with Mass General Brigham affiliate facilities who have undergone an endoscopic primary obesity procedure, an endoscopic bariatric revision procedure, or a bariatric surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2028-05-28 (Estimated); Study Completion 2029-05-28 (Estimated)

PRIMARY OUTCOMES:
Change in weight from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  %TBWL
Change in hypertension from pre-procedure to 10 years using blood pressure measurements | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change of hypertension status by comparing blood pressure measurements (systolic/diastolic mmHg) from baseline.
Change in hypertension from pre-procedure to 10 years using medication dosages | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change of hypertension status by comparing change in dosage (mg) of hypertension medications from baseline.
Change in medication dosage to determine change in diabetes status from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change of diabetes status by comparing change in dosage (mg) of diabetes medications from baseline to 10 years.
Change percent value of HgA1c to determine change in diabetes status from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change of HgA1c (%) by comparing lab values from baseline through 10 years.
Change in total cholesterol lab values (mg/dL) from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change in total cholesterol measurements by comparing followup lab values (mg/dL) to baseline.
Change in low density lipoprotein (LDL) lab values (mg/dL) from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change in LDL measurements by comparing followup lab values (mg/dL) to baseline.
Change in high density lipoprotein (HDL) lab values (mg/dL) from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change in HDL measurements by comparing followup lab values (mg/dL) to baseline.
Change in medication dosage (mg) to determine change in total cholesterol (mg/dL) from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change in total cholesterol measurements by comparing change in dosage of cholesterol medications (mg) from baseline to 10 years.
Change in medication dosage (mg) to determine change in High Density Lipoprotein (HDL) (mg/dL) from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change in HDL measurements by comparing change in dosage of cholesterol medications (mg) from baseline to 10 years.
Change in medication dosage (mg) to determine change in Low Density Lipoprotein (LDL) (mg/dL) from pre-procedure to 10 years | Baseline, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change in LDL measurements by comparing change in dosage of cholesterol medications (mg) from baseline to 10 years.
Change in rate of adverse events from procedure to 10 years | Procedure, 1 month, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change in rate of adverse events post-procedure through 10 years
Change in comorbidity medication dosages from baseline to 10 years | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Change of dosage of comorbidity medications compared to baseline

SECONDARY OUTCOMES:
Change in gastric motility from baseline to 10 years | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Gastric emptying breath test
Change in PYY gut hormones from baseline to 10 years | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months, years 1-10.
  PYY lab values will be compared to baseline
Change in GLP1 gut hormones from baseline to 10 years | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months, years 1-10.
  GLP1 lab values will be compared to baseline
Change in ghrelin hormones from baseline to 10 years | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months, years 1-10.
  Ghrelin lab values will be compared to baseline
Cost comparison of procedural costs associated with bariatric endoscopic vs. surgical procedures from baseline to 10 years | Pre-intervention/procedure/surgery, during the procedure/surgery, immediately after the intervention/procedure/surgery, up to 3 months after the intervention/procedure/surgery
  Cost-effectiveness analysis of procedure costs from admission to discharge for endoscopic vs. surgical bariatric procedures

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Thompson, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the range of data and publication status, the PI will consider de-identified data sharing with a data transfer agreement in place after discussion of parameters and study design.

REFERENCES:
- [Background] Abu Dayyeh BK, Bazerbachi F, Vargas EJ, Sharaiha RZ, Thompson CC, Thaemert BC, Teixeira AF, Chapman CG, Kumbhari V, Ujiki MB, Ahrens J, Day C; MERIT Study Group; Galvao Neto M, Zundel N, Wilson EB. Endoscopic sleeve gastroplasty for treatment of class 1 and 2 obesity (MERIT): a prospective, multicentre, randomised trial. Lancet. 2022 Aug 6;400(10350):441-451. doi: 10.1016/S0140-6736(22)01280-6. Epub 2022 Jul 28. PMID 35908555
- [Background] Jirapinyo P, Thompson CC. Endoscopic gastric plication for the treatment of weight regain after Roux-en-Y gastric bypass (with video). Gastrointest Endosc. 2022 Jul;96(1):51-56. doi: 10.1016/j.gie.2022.02.051. Epub 2022 Mar 5. PMID 35259393
- [Background] de Moura DTH, Hirsch BS, Boghossian MB, de Medeiros FS, McCarty TR, Thompson CC, de Moura EGH. Low-cost modified endoscopic vacuum therapy using a triple-lumen tube allows nutrition and drainage for treatment of an early post-bariatric surgery leak. Endoscopy. 2022 Jul;54(7):E376-E377. doi: 10.1055/a-1540-5870. Epub 2021 Aug 9. No abstract available. PMID 34374043
- [Background] de Moura DTH, de Freitas Junior JR, de Souza GMV, de Oliveira GHP, McCarty TR, Thompson CC, de Moura EGH. Endoscopic management of acute leak after sleeve gastrectomy: principles and techniques. Endoscopy. 2022 Jul;54(7):E327-E328. doi: 10.1055/a-1525-1661. Epub 2021 Jul 9. No abstract available. PMID 34243196
- [Background] Sanchez-Luna SA, Thompson CC, De Moura EGH, de Medeiros FS, De Moura DTH. Modified endoscopic vacuum therapy: Are we ready for prime time? Gastrointest Endosc. 2022 Jun;95(6):1281-1282. doi: 10.1016/j.gie.2021.12.049. No abstract available. PMID 35589208
- [Background] Bazarbashi AN, Dolan RD, McCarty TR, Jirapinyo P, Thompson CC. Endoscopic revision of gastrojejunal anastomosis for the treatment of dumping syndrome in patients with Roux-en-Y gastric bypass: a systematic review and meta-analysis. Surg Endosc. 2022 Jun;36(6):4099-4107. doi: 10.1007/s00464-021-08731-4. Epub 2021 Oct 20. PMID 34669046
- [Background] Jirapinyo P, Thompson CC. Primary Bariatric Procedures. Dig Dis Sci. 2022 May;67(5):1674-1687. doi: 10.1007/s10620-022-07393-z. Epub 2022 Mar 29. PMID 35348970
- [Background] Argueta PP, Salazar M, Vargo JJ, Chahal P, Rodriguez JJ, Simons-Linares CR, Thompson CC. Thirty-Day Readmission After Bariatric Surgery: Causes, Effects on Outcomes, and Predictors. Dig Dis Sci. 2022 Mar;67(3):834-843. doi: 10.1007/s10620-021-06934-2. Epub 2021 Jun 24. PMID 34169433
- [Background] Jirapinyo P, McCarty TR, Dolan RD, Shah R, Thompson CC. Effect of Endoscopic Bariatric and Metabolic Therapies on Nonalcoholic Fatty Liver Disease: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2022 Mar;20(3):511-524.e1. doi: 10.1016/j.cgh.2021.03.017. Epub 2021 Mar 13. PMID 33727164
- [Background] Singh S, Bazarbashi AN, Khan A, Chowdhry M, Bilal M, de Moura DTH, Jirapinyo P, Thakkar S, Thompson CC. Primary obesity surgery endoluminal (POSE) for the treatment of obesity: a systematic review and meta-analysis. Surg Endosc. 2022 Jan;36(1):252-266. doi: 10.1007/s00464-020-08267-z. Epub 2021 Feb 1. PMID 33523277
- [Result] Thompson CC, Jirapinyo P, Shah R, Simsek C. Gastroplasty With Endoscopic Myotomy (GEM) for the Treatment of Obesity: Preliminary Efficacy and Physiologic Results. Gastroenterology. 2022 Nov;163(5):1173-1175. doi: 10.1053/j.gastro.2022.07.077. Epub 2022 Aug 10. No abstract available. PMID 35961376
- [Result] Jirapinyo P, Thompson CC. Comparison of distal primary obesity surgery endolumenal techniques for the treatment of obesity (with videos). Gastrointest Endosc. 2022 Sep;96(3):479-486. doi: 10.1016/j.gie.2022.04.1346. Epub 2022 May 11. PMID 35568242